CLINICAL TRIAL: NCT06142851
Title: Management of Women With Superficial Dyspareunia
Acronym: dyspareunie
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_017_PEC-dyspareunie
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Superficial Dyspareunia
Keywords: superficial dyspareunia; management
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with superficial dyspareunia: Adult women, having sexual activity with or without vaginal penetration, suffering from superficial dyspareunia, whether or not managed by health professionals.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — data collection

SUMMARY:
Superficial dyspareunia are persistent or recurrent pains during an attempt at sexual intercourse or during effective penetration.

They affect between 3 to 18% of women and are a source of physical and psychological suffering.

Some health professionals (gynecologists, general practitioners, midwives) are confronted daily with these complaints.

The approach of sexuality remains a complex subject even within the medical field. As a result, communication between women and health professionals can be difficult, leading to delayed diagnosis or inadequate management.

DETAILED DESCRIPTION:
The main objective is to describe the management of superficial dyspareunia by health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Superficial dyspareunia, i.e.:

  * Having already had several painful vaginal penetrative sex
  * Having pain at the intromission (at the beginning of the vagina and at the level of the vulva) and/or at the beginning of penetration (by a penis, fingers, sextoys)
  * Having persistent and/or recurrent pain (appearing in a manner regular)
* Agreeing to participate in the study

Exclusion Criteria:

* Minors
* Protected by law (guardianship, curatorship, safeguarding of justice)
* Refusing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with superficial dyspareunia
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
medical history | Day 0
  Question to the woman about possible pain during sexual intercourses by an health professional (yes or no)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ufr Medecine Urca, Reims
  - Université de Reims Champagne Ardenne, Reims

IPD SHARING:
Plan to Share IPD: Undecided